CLINICAL TRIAL: NCT02982720
Title: A Phase II Multi-center Study Evaluating Combination Immunotherapy for Advanced Cholangiocarcinoma With Pembrolizumab and Sylatron (Peginterferon Alfa-2b) HCRN:GI16-263
Brief Title: Evaluating Combination Immunotherapy for Advanced Cholangiocarcinoma With Pembrolizumab and PEG-Intron
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Manufacturer discontinued Sylatron
Sponsor: Aiwu Ruth He, MD (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Roswell Park Cancer Institute (Other); The Cleveland Clinic (Other); Georgetown University (Other); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Aiwu Ruth He, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GI16-263
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Results first posted 2019-06-05 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Advanced Cholangiocarcinoma
Keywords: cholangiocarcinoma; Pembrolizumab; MK-3475; Sylatron; peginterferon alfa-2b
MeSH Terms: conditions — Cholangiocarcinoma | interventions — pembrolizumab; peginterferon alfa-2b

STUDY DESIGN:
Masking Description: Open-Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab and Sylatron (Experimental): Pembrolizumab will be administered intravenously at a dose of 200 mg every 3 weeks starting week 4. Sylatron will be administered at a dose of 200mcg subcutaneously weekly starting at week 1.
  Interventions: Drug: Pembrolizumab; Drug: Sylatron

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be administered intravenously.
  Other Names: MK-3475
Drug: Sylatron — Sylatron will be administered subcutaneously.
  Other Names: Peginterferon alfa-2b

SUMMARY:
This is an open-label, single-arm, multicenter Phase II safety and efficacy study of combination therapy with pembrolizumab and Sylatron (Peginterferon alpha-2b) in patients with advanced cholangiocarcinoma who have progressed on or cannot tolerate frontline chemotherapy.

DETAILED DESCRIPTION:
Pembrolizumab and Sylatron Administration:

Pembrolizumab has been evaluated at 2 mg/kg every 3 weeks (Q3W), 10 mg/kg Q3W, or 10 mg/kg Q2W in multiple previous studies for different types of cancer, the response rate at higher dose level seems not improved compared to that of lower dose level. With concerns of increased toxicities from the combination pembrolizumab and sylatron therapy, the pembrolizumab dose is selected to be 200mg administered every three weeks. The approved dose of sylatron for melanoma is induction treatment at 6 μg/kg/week for 8 doses followed by 5 year of maintenance treatment at 3 μg/kg/week for up to 5 years. The approved dose of sylatron for chronic hepatitis C infection in combination with ribavirin is 1.5μg/kg weekly for 24 to 48 weeks.

Each cycle = 21 days or 3 weeks. Based on the approved dosage of sylatron, we decided to treat patients at 200mcg weekly up to 12 weeks (3 weeks as single agent, and 9 weeks in combination of pembrolizumab). Sylatron will start Cycle 1 Day 1 and continue on a weekly basis. We have prepared to reduce the dose of sylatron to 120mcg weekly, or 60mcg weekly if patients experience unacceptable toxicities at the higher dose level of sylatron.

Pembrolizumab will be administered intravenously as a 30 minute infusion at a dose of 200 mg every 3 weeks starting Week 4. Pembrolizumab will start Cycle 2 Day 1 and continue every 3 weeks. All trial treatments will be administered on an outpatient basis.

Sites should make every effort to target infusion timing to be as close to 30 minutes as possible. However, given the variability of infusion pumps from site to site, a window of -5 minutes and +10 minutes is permitted (i.e., infusion time is 30 minutes: -5 min/+10 min).

With concerns about toxicity while using long-term sylatron, if no additional benefit is seen beyond 12 weeks of treatment on top of that expected from pembrolizumab alone, patients will discontinue sylatron treatment after they have received 12 weeks of this therapy (3 weeks as single agent and 9 weeks in combination with pembrolizumab). Pembrolizumab should be continued in the absence of unacceptable toxicity (based on CTCAE v4) until disease progression-based on RECIST 1.1. In patients who had responded to the combination therapy, when patient shows disease progression while on single agent pembrolizumab treatment, Sylatron may be resumed at the discretion of the site investigator after discussion with the sponsor-investigator.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be at least 18 years of age on day of signing informed consent.
3. Patients must have received 1 line of prior systemic therapy for metastatic or resectable disease (i.e. patients may have received adjuvant gemcitabine and then later gemcitabine/cisplatin for recurrent metastatic disease)
4. Histological confirmation of cholangiocarcinoma.
5. Have measurable disease based on RECIST 1.1.
6. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the sponsor-investigator.
7. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
8. Demonstrate adequate organ function:

   Hematological:
   * Absolute neutrophil count (ANC) ≥ 1,500 /μL
   * Platelets ≥ 100,000 / μL
   * Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)

   Renal:
   * Serum creatinine OR Measured or calculated creatinine clearance ≤ 1.5 X upper limit of normal (ULN) OR ≥ 60 mL/min for subject with creatinine levels
   * (GFR can also be used in place of creatinine or CrCl) > 1.5 x institutional ULN

   Hepatic:
   * Serum total bilirubin ≤ 2.0 X ULN
   * AST (SGOT) and ALT (SGPT) ≤ 3.0 X ULN OR ≤ 5 X ULN for subjects with liver metastases
   * Albumin > 2.5 mg/dL

   Coagulation:
   * International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
   * Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential should be willing to use adequate birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
11. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

1. A history of anaphylaxis to peginterferon alfa-2b or interferon alfa-2b
2. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has a known history of active Bacillus Tuberculosis (TB)
5. Hypersensitivity to pembrolizumab or any of its excipients.
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has known history of, or any evidence of active, non-infectious pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the site investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B without HBV treatment (HBV infection with ongoing HBV treatment is allowed); has persistent chronic Hepatitis C infection (successfully treated HCV infection is allowed).
19. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
20. Has history of bipolar disorder or major depression.
21. Has history of not tolerating interferon treatment.
22. Has known serious neuropsychiatric condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2018-02-09 (Actual); Study Completion 2018-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aiwu R. He, MD PhD, Study Chair — Lombardi Comprehensive Cancer Center Georgetown University
Locations (1):
- Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Hoosier Cancer Research Network Website — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab and Sylatron
Started | 4
Completed | 0
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab and Sylatron
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Age, Continuous [Median (Full Range); unit: years] | 66.5 [64 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 4
Disease Subtype [Count of Participants; unit: Participants]
  Extrahepatic | 1
  Gallbladder | 0
  Hilum | 0
  Intrahepatic | 3

OUTCOME MEASURES:

1. Primary Outcome: Asses Objective Response Rate (ORR) of All Patients Receiving Pembrolizumab and Sylatron Combination Therapy
Description: Defined as the proportion of subjects who achieve the best response (CR and PR) determined by RECIST1.1
Time Frame: 12 months
Population: No data was collected or analyzed for this objective due to the early termination of the study by the funder.
Arm/Group | Pembrolizumab and Sylatron
Number analyzed (Participants) | 0

2. Secondary Outcome: Assess Progression Free Survival (PFS) of Patients Receiving Pembrolizumab and Sylatron
Description: Defined as time from start of the treatment till the patient's disease progression or death from any cause (those for whom event of progression or death not observed will be censored).
Time Frame: 36 months
Population: No data was collected or analyzed for this objective due to the early termination of the study by the funder.
Arm/Group | Pembrolizumab and Sylatron
Number analyzed (Participants) | 0

3. Secondary Outcome: Asses Overall Survival (OS) of Patients Receiving Pembrolizumab and Sylatron
Description: Defined as time from start of the treatment till the patient's death from any cause (patient who are still alive at the end of the study will be censored).
Time Frame: 36 months
Population: No data was collected or analyzed for this objective due to the early termination of the study by the funder.
Arm/Group | Pembrolizumab and Sylatron
Number analyzed (Participants) | 0

4. Secondary Outcome: Assess Objective Response Rate (ORR)
Description: the sum of complete response (CR) + confirmed partial response (PR) and will be determined as per irRC.
Time Frame: 36 months
Population: No data was collected or analyzed for this objective due to the early termination of the study by the funder.
Arm/Group | Pembrolizumab and Sylatron
Number analyzed (Participants) | 0

5. Secondary Outcome: Assess Adverse Events, Serious Adverse Events and Serious Adverse Events Leading to Discontinuation of the Treatment (Death) of Combined Pembrolizumab and Sylatron Therapy.
Description: the combination of Sylatron and pembrolizumab as assessed by CTCAE v4
Time Frame: 36 months
Population: No data was collected or analyzed for this objective due to the early termination of the study by the funder.
Arm/Group | Pembrolizumab and Sylatron
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Pembrolizumab and Sylatron
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 4/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab and Sylatron (N=4)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1)
FEVER (General disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab and Sylatron (N=4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (3)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 (6)
ANEMIA (Blood and lymphatic system disorders) | 2 (2)
ANOREXIA (Metabolism and nutrition disorders) | 1 (1)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 (5)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (2)
BLURRED VISION (Eye disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 1 (1)
ENDOCRINE DISORDERS (Endocrine disorders) | 1 (1)
FATIGUE (General disorders) | 4 (4)
GLAUCOMA (Eye disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 3 (5)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 1 (2)
NAUSEA (Gastrointestinal disorders) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1)
PAIN (General disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 1 (1)
WHITE BLOOD CELL DECREASED (Investigations) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated by the funder due to the discontinuation of Sylatron.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT02982720/Prot_SAP_000.pdf